## **INFORMED CONSENT FORM**

Determination of factors affecting early mobilization of patients who have undergone

knee and hip arthroplasty

**Document date:** 08/06/2020

NTC Number: No



## BURSA ULUDAG UNIVERSITY HEALTH SCIENCES RESEARCH AND PUBLISHING ETHICS COMMITTEE RESEARCH APPLICATION FORM

FR 3.8.2 05

(Postscript 5-5)

## BURSA ULUDAG UNIVERSITY HEALTH SCIENCES RESEARCH AND PUBLISHING ETHICS COMMITTEE INFORMED VOLUNTEER FORM FOR SURVEY RESEARCH

Please take time to read this document carefully.

We invite you to a research based on the survey titled "Determination of factors affecting early mobilization of patients who have undergone knee and hip arthroplasty" conducted by Akif BULUT and Nursel VATANSEVER. Before deciding whether to participate in this research or not, you need to know why and how the research will be conducted. For this reason, it is very important to read and understand this form. Take time to carefully read the information below. If you wish, discuss this information with your family and / or relatives. If there are things you do not understand and are not clear to you, or if you want more information, ask us.

Participation in this survey study is completely <u>voluntary</u>. You have the right not to participate in the study. <u>Your response to the questionnaire will be interpreted as giving your consent to participate in the research.</u> Do not be under the pressure or suggestion of anyone while answering the questions on the questionnaires provided to you. The information obtained from these forms will be used purely for research purposes.

This questionnaire consists of 60 questions and takes approximately 20 minutes.

Research Supervisor

Nursel VATANSEVER

**Assistant Professor** 

First Publication Date: 08.06.2020 Revision No / Date: 0 Page 4/10

The latest version published on our website is a controlled document.

**Date of Approval:** 03/10/2017.